CLINICAL TRIAL: NCT03468166
Title: Data Collection for Motor Function and Gait Pattern Analysis of Patients With Chronic Stroke
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-02-053
Record Dates: First submitted 2018-03-06; First posted 2018-03-16 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2019-09

CONDITIONS: Chronic Stroke
Keywords: Motor function; Gait pattern

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic stroke: The data for motor function and gait pattern analysis was obtained.
  Interventions: Other: Chronic stroke

INTERVENTIONS:
Other: Chronic stroke — The data for motor function and gait pattern analysis was obtained.

SUMMARY:
In chronic stroke patients, the data for motor function and gait pattern analysis was obtained.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients with hemiplegia over 19 years old
* Ischemic or hemorrhagic stroke patients over 6 months of onset
* Functional Ambulation Category Scale with 3 or more scales and a person who can walk independently regardless of using of walking aids
* A person who understands and voluntarily participates in this study and signs a research agreement

Exclusion Criteria:

* Patients of artificial heartbeat
* Patients with claustrophobia
* Patients with intracranial metal implants
* Patients who are contraindicated for other common MRI scans
* Patients difficult to walk due to problems such as visual field defect, fracture, severe muscle paralysis, cognitive impairment
* Those who have a score of FMA score of 80 or more and have very slight motor impairment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with chronic stroke who can walk outdoors
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Gait analysis | 1 hour
  Gait analysis is a process of measuring and evaluating the walking patterns of patients by using surface electromyograph and motion analysis system.

SECONDARY OUTCOMES:
Fugl-Meyer assessment for lower extremity (FMA) | 20 minutes
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment.
The Timed Up and Go test (TUG) | 10 minutes
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
10 meter walk test (10MWT) | 5 minutes
  Measure of self selected speeds by measuring the time it takes an individual to walk 10 meters. To perform the test, patient walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: "Please walk this distance at your normal pace when I say go."
Manual Muscle Test (MMT) | 15 minutes
  Manual muscle testing (MMT) is a procedure for the evaluation of the function and strength of individual muscles and muscle groups based on the effective performance of a movement in relation to the forces of gravity and manual resistance.
Range of Motion (ROM) | 15 minutes
  Range of Motion (ROM) testing is the measurement of movement around a specific joint or body part.
Functional Ambulation Classification (FAC) | 10 minutes
  The Functional Ambulation Categories (FAC) is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device.
Modified Bathel index (MBI) | 10 minutes
  The MBI is a measure of activities of daily living, which shows the degree of independence of a patient from any assistance. It covers 10 domains of functioning (activities): bowel control, bladder control, as well as help with grooming, toilet use, feeding, transfers, walking, dressing, climbing stairs, and bathing.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea